CLINICAL TRIAL: NCT04408534
Title: Bilevel Noninvasive Ventilation in Infants With Bronchiolitis Presenting With Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A01183-36
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-04

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous positive airway pressure (Active Comparator): Patients receive continuous positive airway pressure as a mode of noninvasive ventilation
  Interventions: Other: mode of noninvasive ventilation
- bilevel positive airway pressure (Experimental): Patients receive bilevel positive airway pressure as a mode of noninvasive ventilation
  Interventions: Other: mode of noninvasive ventilation

INTERVENTIONS:
Other: mode of noninvasive ventilation — administration of during 3 hours each 4 cycles

SUMMARY:
This physiological study aims to compare Bilevel Positive Airway Pressure and continuons positive airway pressure in infants with severe bronchiolitis presenting with apnea

DETAILED DESCRIPTION:
This study is a cross over randomized study which aims to compare the effect of 2 modes of noninvasive ventilation on the occurence of central apnea, as measured by electrical activity of the diaphragm

ELIGIBILITY:
Inclusion Criteria:

* Children born at gestational age > 36 weeks gestation
* Ventilated in Non Invasive Ventilation (NIV) for acute bronchiolitis (clinical criteria of the American Academy of Pediatrics)
* Having presented at least 1 apnea objectified by the parents or by a health care professional, as previously described (1), with one or more of the following characteristics: 1/Associated with bradycardia < 80 / min, 2/Associated with desaturation < 85% or 3/Duration more than 10 seconds
* Informed consent signed by at least one of the two parents + oral agreement from the second parent before the intervention of the study (2nd signature to be collected as soon as possible)

Exclusion Criteria:

* With chronic respiratory insufficiency requiring home ventilation (NIV or under long-term oxygen therapy, initiated at least 14 days before the start of the study)
* Ventilated in NIV for more than 48 hours before inclusion
* Hemodynamically significant cardiac disease, primary ENT or pulmonary pathology (malformative or genetic) or neuromuscular pathology
* Presenting a contraindication of a gastric tube (trauma or recent surgery concerning the cervical, pharyngeal or esophageal regions, severe coagulation disorders)
* Patient not affiliated to health care insurance

Ages: 3 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Apnea | Up to 12 hours
  Number of apnea

IPD SHARING:
Plan to Share IPD: Undecided